CLINICAL TRIAL: NCT04629235
Title: Reduction of Bedrest Time of Post Percutaneous Renal Biopsy Patients (RBP) Evaluated by Nursing Outcomes Classification (NOC): a Randomized Clinical Trial
Brief Title: Reduction of Bedrest Time of Post Percutaneous Renal Biopsy Patients
Acronym: RUBBY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 170430
Record Dates: First submitted 2020-10-30; First posted 2020-11-16 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Bedrest
Keywords: Renal Biopsy; Complications; Standardized Nursing Terminology
MeSH Terms: interventions — Bed Rest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24 hours of bedrest (Active Comparator): - 24 hours of bedrest
  Interventions: Behavioral: bedrest
- Intervention group (Experimental): - Wonder around after 8 hours of bedrest
  Interventions: Other: wonder around

INTERVENTIONS:
Other: wonder around — wonder around after 8 hours of bedrest
  Arms: Intervention group
Behavioral: bedrest — 24 hours of bedrest
  Arms: 24 hours of bedrest

SUMMARY:
To compare the reduction of the bedrest time of the patient after percutaneous renal biopsy from 24 hours to 8 hours in relation to the occurrence of complications evaluated by the Nursing Outcome Classification (NOC) indicators.

DETAILED DESCRIPTION:
Percutaneous renal biopsy (BRP) is an important procedure for the diagnosis, prognostic evaluation and therapeutic orientation of several kidney diseases. Although it is considered a safe procedure, BRP complications can occur and, most of the time, are related to the risk of bleeding and the main consequence of BRP. Complications include macroscopic hematuria and hematoma requiring blood transfusion, surgical intervention, or invasive procedure. Since hemorrhagic complications continue to be the highest risk after BRP due to severity and potential life-threatening risk, there is an effort to minimize the risk of bleeding by checking blood clotting markers prior to the procedure, uncontrolled hypertension and the use of antiplatelet drugs and anticoagulants. The relevance of this study is to seek better evidence for clinical practice, considering the lack of Brazilian studies on the subject and the positive impact on patient comfort, besides the reduction of costs for the institution and overload in the work of the multidisciplinary team. In addition, it will contribute to the strengthening of the use of NOC in clinical practice and to the improvement of nursing knowledge.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing renal biopsy at Hospital de Clínicas de Porto Alegre (HCPA);
* Both sexes;
* Aged 18 years or older.

Exclusion Criteria:

* Patients with the following risk factors for complications;
* More than two punctures during the procedure;
* Larger gauge needle;
* Uncontrolled blood pressure;
* Blood clotting disorders and use of antiplatelet agents (aspirin or clopidogrel), or use of anticoagulants;
* Bedridden patients and patients unable to adequately to ambulate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
NOC Blood coagulation (0409) | 24 hours
  The primary outcome will be constituted of the absence of bleeding, measured according to the clinical indicators Bleeding (040902), Bruising (040903) and Hematuria (040918). Checked by visual inspection at the puncture location. Check hematuria by visual inspection and test with reagent strips. Evaluated by Likert scale, being 1 the worst score and 5 best score.
  NOC Blood loss severity (0413): Meansurement of indicators Abdominal distension (041306) and Skin and mucous membrane pallor (041313). Assess the abdominal distension of the patient in the supine position, through inspection and palpation. Assess pallor by inspecting the extremities and mucous membranes, associated with the evaluation of capillary filling with the compression/decompression of the pulp of one or more digits. Evaluated by Likert scale, being 1 the worst score and 5 best score.

SECONDARY OUTCOMES:
NOC Circulation status (0401) | 24 hours
  Measurement of Systolic blood pressure (040101) and Diastolic blood pressure (040102) with an inflatable cuff. Evaluated by Likert scale, being 1 the worst score and 5 best score.
NOC Pain level (2102) as assessed by Visual Analog Pain Scale or Numerical Verbal Pain Scale, asking how much they rate their pain from 0 to 10 | 24 hours
  The improvement of the indicators Reported pain (210201) and Facial expressions of pain (210206). Question the patient about their pain level using a Visual Analog Pain Scale or Numerical Verbal Pain Scale, asking how much they rate their pain from 0 to 10. Evaluated by Likert scale, being 1 the worst score and 5 best score.
NOC Comfort status: physical (2010) | 24 hours
  Maintenance of Physical well-being (201002) and Comfortable position (201004). Question the patient about physical well-being and see if he has characteristics, for example: good physical mobility; feels comfortable; normal breathing; absence or control of pain. Ask the patient if he is comfortable with his body position. Check the need to use non-pharmacological (pillow, cushion, etc.) and/or pharmacological methods to be able to position yourself comfortably. Evaluated by Likert scale, being 1 the worst score and 5 best score.

CONTACTS AND LOCATIONS:
Overall Officials: Amália de Fátima Lucena, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No